# **Detailed Protocol: Denosumab and High-dose Teriparatide Administration Study (DATA 2)**

## I. Background and Significance

As our population ages, osteoporotic fractures are expected to have an increasing impact on the health of our population. Today, osteoporosis is estimated to affect over 20 million Americans with 1.5 million osteoporotic fractures occurring in the United States every year <sup>1</sup>. In women, the lifetime risk of experiencing a minimal trauma hip fracture, the most devastating consequence of osteoporosis, is estimated to be 17% 2. In most patients with osteoporosis, the occurrence of a hip fracture is a devastating consequence, conveying 24% excess mortality within 12-months of the fracture and a continued increased risk of death for up to 10-years after the event 3. In patients with the most advanced osteoporosis, currently available medications can, at best, decrease hip and non-spine fracture rates by 50% and 30%, respectively <sup>4,5</sup>. At present, the mainstay of osteoporosis treatment is the use of oral and intravenous bisphosphonates (BPs). These drugs act by suppressing bone resorption (as well as formation) and have been shown to increase bone mineral density (BMD) and reduce fracture rates in certain populations <sup>6</sup>. Teriparatide (TPTD- hPTH 1-34) has also been shown to increase BMD and reduce fractures, but acts by a different mechanism that involves stimulating new bone formation (along with resorption), and reconstituting internal bone microarchitecture 7-14. The effects of TPTD are dose dependant both with regard to increases in bone mass and stimulation of osteoblast activity <sup>13</sup>. Specifically, biochemical markers of bone formation increase more in women treated with 40-µg of TPTD daily compared to women treated with 20-µg (the FDA approved dose) and this greater stimulation of bone formation is associated with greater BMD increases, particularly in trabecular bone 14,15. Despite stimulating greater increases in bone mass, TPTD 40 mcg/day reduces spine and non-spine fractures no more than TPTD 20 mcg/day in humans. We hypothesize that this paradox arises because 40-mcg/day increases bone resorption more than 20-mcg/day, a difference revealed by biochemical markers of bone resorption <sup>14,16</sup>. Unique among osteoporosis medications, TPTD has also been shown to stimulate periosteal expansion in animal models though a similar property in human studies has yet to be unequivocally shown 8,17-19.

While both TPTD and BPs increase BMD and reduce fracture risk, their beneficial effects are limited and neither drug is able to completely normalize BMD or restore skeletal integrity in most patients. Initially thought to be a promising approach, trials of combination therapy with anabolic agents and BPs have demonstrated minimal or no advantage over monotherapy <sup>20-26</sup>. In these combination studies, the antiresorptive agent inhibited TPTD or PTH-stimulated increases in bone formation and resorption but did not suppress turnover to the degree observed with the antiresorptive agent alone <sup>22-26</sup>. Together, these studies suggest that co-administration of BPs with TPTD blunts the TPTD-associated stimulation of bone formation in a dose-dependent fashion, particularly in predominately trabecular sites such as the spine. The reasons that the combination of BPs and TPTD do not stimulate greater gains in BMD are unclear. BPs presumably interfere with one or more of the mechanisms via which TPTD exerts its anabolic effect on bone: increased secretion of IGF-I, bFGF, or other paracrine growth factors by osteoblasts, decreased production of sclerostin by osteocytes, and/or increased osteoclastic resorption of bone with resultant release of these and other pre-formed growth factors <sup>23,27,28</sup>.

Rodent models have suggested that TPTD in combination with OPG (a molecule aimed at the same molecular target as denosumab— see below) has superior skeletal effects compared to TPTD alone <sup>29,30</sup>. Denosumab (DMAB) is an FDA-approved fully human monoclonal antibody that specifically binds to receptor activator of nuclear factor-kB ligand (RANKL)<sup>31</sup>. It inhibits bone resorption by interfering with the binding of RANKL to its receptor on pre-osteoclasts and osteoclasts, the final common pathway leading to osteoclast activation and bone resorption <sup>32,33</sup>. DMAB suppresses bone turnover more than intravenous and oral BPs <sup>34,35</sup>. DMAB's potent antiresorptive properties are best demonstrated in iliac crest biopsy specimens from postmenopausal osteoporotic women who had been taking the drug for 24-36 months. These biopsies revealed an 80% reduction in eroded surface

and the complete absence of osteoclasts in more than 50% of the specimens. Furthermore, histomorphometric indices of bone turnover were significantly lower in the patients taking DMAB than those taking alendronate <sup>36</sup>. Despite this dramatic suppression of osteoclast activity, however, bone turnover rapidly normalizes after the drug is discontinued <sup>31</sup>. Like other antiresorptive agents, DMAB increases BMD at the lumbar spine and hip, but unlike most of these agents also increases BMD at diaphyseal sites such as the wrist <sup>37-42</sup>. Furthermore, DMAB reduces the risk of vertebral and hip fractures in postmenopausal women with osteoporosis, and increases indices of bone strength when measured by HR-pQCT <sup>43,44</sup>. Taken together, the unique mechanism of action of DMAB and the suggestive animal studies led us to hypothesize that the combination of DMAB and TPTD would increase BMD, bone guality, and estimated bone strength more than either drug alone.

This hypothesis was tested and confirmed in The DATA Study (ClinicalTrials.gov Identifier NCT00926380) <sup>45,46</sup> that compared teriparatide and denosumab monotherapy to the combination of both drugs in postmenopausal osteoporotic women. As shown below, the results not only showed that the combination increased hip and spine BMD more than either drug alone, but also that in the presence of DMAB, the pro-resorptive effects of TPTD are completely blocked (unlike combinations of TPTD and BPs).



The combination group is statistically different from both other groups at all sites (P<0.02). TPTD group is statistically different from DMAB at total hip only



For clarity, changes are shown for combination and DMAB groups only (\*P=0.05 for between-group comparison). In the TPTD alone group, typical increases in OC, P1NP (bone formation markers), and CTX (bone resorption marker) were observed.

These results suggest that even greater gains in BMD, bone quality, and bone strength could be achieved if DMAB could be combined with a more potent stimulant of osteoblast function and bone formation. Thus, we plan to conduct 15-month study that compares TPTD 40-µg plus DMAB (60-mg every six months) to TPTD 20-µg plus DMAB in a design that also takes advantage of recent work that suggests that starting TPTD before the antiresorptive has some clinical advantages <sup>47,48</sup>.

In performing this clinical trial, we will be able to better understand the mechanisms by which antiresorptive agents influence the efficacy of anabolic agents. Furthermore, if our hypothesis is confirmed, the findings of this study could define a novel approach to the treatment of high-risk osteoporosis patients.

A known limitation of both teriparatide and denosumab therapy is the rapid loss of bone that occurs when these drugs are discontinued. 49,50 Moreover, both teriparatide and denosumab are expensive and administered by subcutaneous injection (daily and every 6-months, respectively). If combination teriparatide/denosumab therapy is to become part of a widely used treatment approach, we must develop strategies to maintain and expand the unprecedented improvement in bone density and microarchitrecture observed, and do so with acceptable risk of serious adverse effects. Zoledronic acid is a highly potent bisphosphonate that has been shown to reduce the risk of both vertebral and non-vertebral fractures when given as a yearly 5-mg infusion over 3 years. Despite the FDA-approved yearly dosing schedule, it has also been reported that the effects of a single 5-mg zoledronic acid infusion are much more prolonged. Specifically, a single administration of zoledronic acid continues to reduce bone resorption and increase BMD for an additional 2-5 years. 452-55 Moreover, it has also been demonstrated that a single dose of zoledronic acid continues to reduce fracture rates for at least 3-years and to the same degree as do yearly infusions.

As the optimal treatment for patients who have previously received combination denosumab and teriparatide is not defined, we believe that is useful and important to look at how our study subjects' bone mineral densities have changed a year or more after completion of their participation in our study.

# **II. Specific Aims**

# The Specific Aim of this protocol is to test the following hypothesis:

In postmenopausal women with osteoporosis, the combination of DMAB and high-dose TPTD (which will be started 3-months prior to denosumab) will increase BMD, improve bone microarchitecture, and increase estimated bone strength more than the combination of DMAB and standard dose TPTD.

#### The Specific Aim of the Extension trial (DATA-2-EX):

The extension trial described (DATA-2-EX) will test the hypothesis that the large increases in cortical and trabecular BMD, bone quality, and estimated bone strength achieved with combined DMAB and high-dose TPTD therapy can be extended for up to 27-months by a single 5-mg dose of zoledronic acid. If this hypothesis is confirmed, it will represent a significant advance in the rational development of comprehensive treatment strategies, especially for those with severe disease in whom single-agent therapy does not adequately reduce fracture risk. Additionally, positive results from DATA-2-EX would support the initiation of a larger trial assessing the anti-fracture efficacy of this approach.

#### The Specific Aim of the Observational visit:

This optional observational visit is specific to subjects who completed the month-15 trial but did not enroll in DATA-2-EX. We wish to test the hypothesis that further transitioning to intravenous bisphosphonate from the two treatment groups will prevent the bone loss associated with discontinuing these therapies and will further increase bone density.

# III. Subject Selection

350 female volunteers will be screened and 70 female volunteers will be recruited by advertisement in accord with institutional guidelines for clinical studies. Recruitment flyers will be posted in approved locations throughout the MGH (including the MGH Bone Mineral Density Center) and email announcements will be sent through the Partners Clinical Research Program Network. Letters will be sent to subjects identified through RSVP for Health. Additionally, advertisements will be published in local newspapers and a mailing will be sent to targeted populations, including subjects who have expressed an interest in one of our research group's previous studies.

Subjects will be paid \$50 after each completed visit (other than the screening visit) for a total of \$300.

Parking vouchers will be provided to subjects at each visit, including the screening visit.

#### Inclusion Criteria:

Must satisfy A and B and C and D below:

A. women aged > 45

- B. postmenopausal by either of the following criteria:
  - > 36 months since last spontaneous menses;

or

- > 36 months since hysterectomy, plus serum FSH > 40 units / liter.
- C. osteoporosis with high risk of fracture' by one or more of the following criteria:

DXA spine or hip T-score ≤ - 2.5;

10

DXA spine or hip T-score  $\leq$  - 2.0 plus  $\geq$  1 of the following BMD-independent risk factors for fracture: fracture after age 50, parental hip fracture after age 50, prior hyperthyroidism, inability to rise from a chair with one's arms elevated, current tobacco smoker.

or

DXA spine, hip, or forearm T-score  $\leq$  - 1.0 plus  $\geq$  1 adult low-trauma fracture (low-trauma fracture = fracture after no trauma; or fracture after falling  $\leq$  6 inches when stationary or moving slower than a run.

## **Exclusion Criteria:**

- confirmed serum alkaline phosphatase above upper normal limit with no explanation
- liver disease (AST or ALT > 2 x upper normal limit).
- renal disease (serum creatinine > 2.0 mg/dl).
- Hypocalcemia or hypercalcemia (Ca <8.5 mg/dL or >10.5 mg/dL)
- Abnormal blood PTH (intact PTH < 10 pg/mL or > 65 pg/mL)
- serum 25-OH vitamin D < 20 ng/ml
- HCT < 32%.
- history of malignancy (except non-melanoma skin carcinoma) or radiation therapy.
- history of gouty arthritis.
- significant cardiopulmonary disease including unstable coronary artery disease, stage D
  ACC/AHA heart failure or any other condition that the investigator deems may preclude the
  subject from participating safely or completing the protocol procedures.
- major psychiatric disease that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
- excessive alcohol use or substance abuse that in the opinion of the investigator would preclude the subject from providing adequate informed consent or completing the protocol procedures.
- known congenital or acquired bone disease other than osteoporosis (including osteomalacia, hyperparathyroidism, Paget's disease)
- current use or use in the past 6 months of oral bisphosphonate
- current use or use within the past 3 months of estrogens, selective estrogen receptor modulators, or calcitonin.
- Current use or use in the past 6 months of denosumab
- use of oral or parenteral glucocorticoids for more than 14 days within the past 6 months
- any current or previous use of strontium, teriparatide, or any parenteral bisphosphonate.

4

- known sensitivity to mammalian cell-derived drug products.
- known sensitivity to teriparatide or any of its excipients.
- known sensitivity to densoumab or any of its excipients.
- Extensive dental work involving extraction or dental implant within the past 2 months or planned in the upcoming 2 months.

#### DATA-2-EX criteria:

Subjects completing DATA-2 will be offered enrollment in DATA-2-EX if they meet the same entry criteria outlined in DATA-2 with the following exceptions related to fracture risk. Subjects currently enrolled will be offered enrollment in DATA-2-EX by letter and a follow-up phone call at least 2 months prior to their 4<sup>th</sup> study visit. Subjects being recruited will be informed of the optional extension during the screening phone call.

All subjects enrolled in DATA-2 will be eligible for DATA-2-EX or the optional observational visit.

In addition to these DATA-2 criteria, to be enrolled in DATA-2-EX, women will be required to have an estimated GFR  $\geq$ 35 (mL/min), a 25-(OH) Vitamin-D level  $\geq$ 20 (ng/mL), and no known allergy to bisphosphonates. Laboratory testing of Cr, GFR and 25-OH vitamin D will be performed within 3 months of receiving zoledronic acid. The exclusion criteria will remain the same as the original DATA-2 exclusion criteria, as outlined above, with the exception that prior exposure to denosumab and teriparatide as part of the DATA-2 protocol are permitted and renal function criteria will be assessed by estimated GFR (rather than the creatinine level). Zoledronic acid will not be infused if the 25-OH vitamin D level is <20 ng/mL or GFR is <35 mL/min.

## **IV. Subject Enrollment**

This outpatient study will either be conducted at one or more of the following sites: the General Clinical Research Center (GCRC), the Osteoporosis Research Center or the Endocrine Unit Clinical Space (all within the Massachusetts General Hospital.

The general design is a randomized, 2-arm, open label study.

# Groups and Randomization

Subjects will first be screened, and those who appear eligible will have a medical history and interview with a study investigator. Those who remain eligible will be formally accepted into the study by a study investigator, assigned to one of 4 strata based on age (above or below 65) and previous bisphosphonate use (previous use or none) and then randomly assigned within each strata to one of the 2 treatment groups by computer-generated cards. (1:1: ratio). Within each of the four strata, the randomization block size will vary randomly to minimize the predictability of treatment assignments.

The study period lasts 15 months. There will be 35 subjects in each group.

All subjects completing the 15-month DATA-2 trial be offered enrollment in the DATA-2-EX study.

For subjects who do not enroll in DATA-2-EX, subjects may enroll for an optional observational visit. The observational period will start immediately after the DATA-2 study's 15-month visit and will last an additional 12 to 24 months. During that interval, each subject will be contacted by phone.

All subjects will be asked if:

- They continued osteoporosis treatment and if so, with what drug

- They have sustained any new fractures.

We will request that all subjects return for one visit to complete one bone density scan of the spine and hip (by DXA) within 12 to 24 months of the completion of the 15-month study. Informed consent for this visit will be obtained by a research assistant. The DXA will be performed at no cost to the study subjects.



Note: (Optional one-time observational visit for only DXA may occur between month 27 and month 39 for subjects who do not receive zoledronic acid.)

All subjects who report dietary intake of less than 1200mg of calcium daily will be given calcium supplementation (600mg elemental calcium) with Vitamin D (400IU). Subjects with a dietary intake > 1200 mg will receive Vitamin D only.

# V. Study Procedures

# Telephone screening and Screening Visit:

Members of research staff will screen all interested subjects over the telephone. If subjects meet initial criteria and are interested in the study, a member of the study staff will schedule a screening visit wherein the subject will sign a separate "screening only" consent form. This consent form will allow for a blood draw and bone mineral density testing.

Prior to signing this screening only consent form, subjects will be offered the option to speak with a physician investigator if they wish or if they have questions that can't be answered by the RA.

At this visit, bone mineral density of the spine and hip will be obtained and the following will be measured in serum or blood:

- PTH
- 25-(OH) Vitamin D
- Routine chemistries (Calcium, Phosphate, electrolytes, BUN, creatinine, ALT)
- Complete Blood Count
- FSH (if necessary because of prior hysterectomy)

# Visit 1:

If the subject meets the above BMD and laboratory criteria, she will then be scheduled for visit 1. At this visit, a study physician will obtain written informed consent for participation in the complete study. If subjects require more time to consider participating after reading the consent form the screening

visit will not continue. If the subject is ready to sign the consent form, the study physician will then perform a history and physical on her. If all inclusion/exclusion criteria are met, subjects will then continue visit 1 and the subsequent visits.

# Visit 1-6:

These visits will occur at the following times:

Visit 1 (month 0)

Visit 2 (month 3 +/- 2 weeks)

Visit 3 (month 9 +/- 2 weeks)

*Visit 4 (month 15 +6/- 2 weeks)* 

Visit 5 (month 27 +/-2 weeks)

Visit 6 (month 42 +/-2 weeks)

If enrolled in optional observational study, these visits will occur at the following times:

Visit 1 (month 0)

Visit 2 (month 3 +/- 2 weeks)

Visit 3 (month 9 +/- 2 weeks)

Visit 4 (month 15 +/- 2 weeks)

Visit 5 (month 27, up to month 39)\_Visit 5 will consist of obtaining informed consent and DXA hip and spine scan only. A blood draw will not be performed.

Subjects will be seen at MGH prior to 10 a.m. and will be instructed to be fasting, and to skip that day's PTH injection (if any). The following blood/serum tests will be measured:

- Routine chemistries (Calcium, Phosphate, electrolytes, BUN, creatinine, ALT, PTH, 25OH vit D)
- Complete Blood Count
- Serum CTX (pooled assay of de-identified samples at end of study to be analyzed by collaborator Dr. Richard Eastell)
- Serum osteocalcin (pooled assay of de-identified samples at end of study to be analyzed by collaborator Dr. Richard Eastell)
- Serum PINP (pooled assay of de-identified samples at end of study to be analyzed by collaborator Dr. Richard Eastell)

After which the subjects will be given breakfast, and then have the following procedures per table below:

The following procedures are performed at each visit:

| | <u>Screen</u> | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|---|
| <u>Month</u> | | 0 | 3 | 9 | 15 | 27 | 42 |
| Routine and hormonal lab testing | <u>X</u> | <u>X</u> | <u>X</u> | <u>X</u> | <u>X</u> | √_ | √_ |
| History and Physical Exam | X | | | | | | |
| Dispense Medications | | <u>X</u> | <u>X</u> | <u>X</u> | √ | | |
| Bone Turnover Markers | | <u>X</u> | <u>X</u> | <u>X</u> | <u>X</u> | √ | <u>√</u> |
| BMD by DXA of PA spine, hip, and 1/3 distal radius | <u>X</u> | <u>X</u> | X | X | <u>X</u> | √,* | √ |
| HR-pQCT of radius and tibia | | <u>X</u> | X | X | X | √ | √ |
| QCT of the hip and spine | | X | | | X | | |

X = DATA-2 procedures √ = DATA-2-EX procedures \*= observational visit, DXA spine and hip only

After blood sampling, denosumab (sold under the brand name Prolia) will be administered (visits 2 and 3 only). Additionally, at visit 1 subjects will be trained in the use of the teriparatide pen (sold under the brand name Forteo®) and will give themselves the first injection while observed by a member of the study staff. At each visit participants will return their used and unused Forteo® injection pens, so we can estimate and record the unused volume in each pen and thereby estimate her compliance with Forteo® use. All subjects in DATA-2-EX receive a single 5-mg infusion of zoledronic acid at month 15.

Study funds and NIH funding will cover the costs of all study procedures, ancillary medications and the costs of the study drugs if not covered by insurance or the manufacturer.

Note: Any remaining serum samples will be saved and may be used to measure other variables related to bone metabolism at a future time. Samples will be stored with subject code number and date and time of sampling in a locked –80 degree freezer and only approved study personnel will have access to the samples. It is understood that any future use of samples must be reviewed and approved separately by the HRC prior to their use. Personal-Identifying information will be removed before any sample is sent out for analysis to a non-Partners affiliated institution.

Note: The Principal Investigator may end the subject's participation without the subject's consent in order to protect the health of the subject, if the subject is unable to attend to study visits, if the sponsor decides to stop the study, or due to other administrative reasons.

## Interpretation of results and study limitations of the proposed clinical trial:

This 15-month RCT will provide scientifically important and potentially groundbreaking clinically relevant findings. The combination of anabolic therapy with BPs has not been promising but the DATA study demonstrates that DMAB, through its distinct mechanism of action, may prove to be a more effective inhibitor of osteoclast activity in the presence of a potent anabolic stimulus. By increasing the TPTD dose, we hypothesize that we will maintain or improve bone formation rates while resorption remains powerfully inhibited. If the combination of this higher TPTD dose and DMAB increases BMD, improves bone quality, and increase estimated bone strength more than the combination of high-dose TPTD and alendronate and the combination of standard-dose TPTD and DMAB, it will represent a significant step forward in osteoporosis therapy. Additionally, analysis of the QCT and HR-pQCT assessments will potentially confirm the robust effects of DMAB and TPTD co-administration on the cortical compartment of the axial and appendicular skeleton.

## VI. Study Endpoint and Statistical Analysis

The primary endpoint is the change in PA spine BMD (DXA) between treatment groups at 15 months. The method of analysis will be a longitudinal mixed effects ANOVA. This model includes the subject level random intercept, time, fixed treatment effect, and the (group)X(time) interaction term. The inference of the regression coefficient associated with the interaction term (difference in slopes) will determine differences between treatment groups. The model will allow us to include all available partial observations for the non-completers and this approach will provide more valid estimates (with increased efficiency) of the time effects than the last value carried forward method.

# Calculation of Power

For purposes of estimation, we calculated the sample based on a between-group comparison of the mean intra-individual treatment effect over the treatment period for the primary and secondary endpoints based on the our observations of the standard deviation of the 12-month treatment effects observed in the DATA study. We predict that 30 subjects in each group will complete the study. This represents an 86% completion rate, a conservative estimate based on our current withdrawal rate of less than 6% in DATA. With this group size, the table below shows our estimated power calculations using the Hsu (With Best) multiple comparison test at a 5% significance level and assuming 80% power. The Hsu completers-based power analysis is conservative, and the actual analysis will likely attain greater power as the full analysis set can be utilized.

| <u>Parameter</u> | Standard Deviation of 12-month change in subjects receiving combination therapy in DATA. | Minimum detectable difference at a 5% significance level assuming 80% power |
|---|---|---|
| DXA PA Spine (primary endpoint) | 3.8% | 2.5% |
| DXA Fem. Neck | 4.3% | 2.8% |
| DXA Total Hip | 2.8% | 1.9% |
| Distal Radius Total vBMD | 2.2% | 1.5% |
| Distal Radius HR-pQCT Cortical vBMD | 1.5% | 1.0% |
| Distal Radius HR-pQCT Cortical Thickness | 4.5% | 2.9% |
| Distal Tibia Total vBMD | 2.1% | 1.4% |
| Distal Tibia HR-pQCT Cortical vBMD | 1.5% | 1.0% |
| Distal Tibia HR-pQCT Cortical Thickness | 3.1% | 2.4% |
| CTX | 35% | 23% |
| Osteocalcin | 27% | 18% |
| P1NP | 32% | 21% |

These detectable between-group differences are at the lower limit of what is considered clinically important and generally correspond to the between-group difference that we observed in the DATA study.

# VII. Risk and Discomforts

# Denosumab

DMAB is an FDA approved medication used to treat osteoporosis in various populations, including postmenopausal women. More than 13,500 patients have been treated with DMAB in clinical studies, and it is generally well tolerated. In clinical studies, it has been reported that DMAB may uncommonly produce the following side-effects: eczema, serious skin infections, low blood calcium (which can cause tingling in the fingers or around the mouth, muscle cramps, or abnormal heart rate), pain in the joints or extremities, high blood cholesterol, dizziness, cough, difficulty emptying the bladder, and decreased skin sensation. Hypocalcemia has been very rarely reported in absence of renal failure. Osteonecrosis of the jaw has been reported in the oncology clinical trial program in patients treated with DMAB but its relative incidence compared to placebo is unclear. Atypical, low-energy, or low trauma fractures of the femoral shaft have been reported patients who received DMAB. The incidence of atypical femur fractures is not well-defined but appears to be extremely rare. If a study subject presents with thigh or groin pain, she will be immediately evaluated to rule out an incomplete femur fracture.

#### Teriparatide

TPTD is an FDA approved medication used to treat postmenopausal women with osteoporosis who are at high risk of fracture. The most commonly reported side effects of TPTD are overall pain, asthenia, nausea, headache, leg cramps, sinus tachycardia, arthralgia, rhinitis), and dizziness. TPTD can cause transient hypercalcemia, which is generally mild, even with the 40-µg dose <sup>13</sup>. Repeated daily administration of TPTD in high doses to rodents causes dose-dependent osteosclerosis, bony obliteration of the marrow space, and extra-medullary hematopoiesis, followed by osteosarcomas. The relevance of these findings to humans is unclear and will remain so for many years, because osteosarcoma is rare in adults (4 cases/million/year). Eli Lilly and the FDA are monitoring the incidence of osteosarcoma in TPTD treated patients and have not reported a linkage thus far.

The dose of TPTD chosen ( $40-\mu g$ ) is higher than that currently approved by the U.S. Food and Drug Administration ( $20-\mu g$  once daily) but the same as doses used in other clinical studies, including our own. Studies from our group were performed under an IND to Dr Robert Neer (co-investigator) and include the following:

| Study | Population | Total subjects<br>receiving TPTD<br>40-µg SC daily | Duration | Hypercalcemia incidence (24-hrs post-dose) |
|---|---|---|---|---|
| Finkelstein et al.<br>NEJM 2003 <sup>24</sup> | men | 55 | 24 months | <1% |
| Finkelstein et al.<br>JCEM 2010 <sup>23</sup> | postmenopausal women | 62 | 24 months | <2% |

In the largest study of the 40- $\mu$ g dose of teriparatide <sup>13</sup>, 541 women received the 20- $\mu$ g dose and 544 women received the 40- $\mu$ g dose for a mean if 19 months. In this study, both doses were generally well tolerated and differences in side effects between doses were small. Side effects included nausea (40- $\mu$ g 18%, 20- $\mu$ g 8%, placebo 8%), headache (40- $\mu$ g 13%, 20- $\mu$ g 8%, placebo 8%), dizziness (40- $\mu$ g 6%, 20- $\mu$ g 9%, placebo 6%), and leg cramps (40- $\mu$ g 1%, 20- $\mu$ g 3%, placebo 1%). Additionally, the 40- $\mu$ g dose was well-tolerated in a group of 122 postmenopausal women when co-administered with hormone replacement therapy for 24 month <sup>15</sup>.

## Zoledronic Acid

The most common side effects associated with zoledronic acid include flu-like symptoms (e.g., fever, chills, muscle/joint aches) occurring after the infusion. The majority of these symptoms occur within the first 3 days following drug administration and usually resolve within 3 days of onset but resolution can take up to 7-14 days. Taking acetaminophen or ibuprofen after the infusion can mitigate these symptoms. Other common side effects include nausea, tiredness, dizziness, headache, or pain/redness/swelling at the injection site.

Renal toxicity: Zoledronic acid, has been associated with renal impairment and in rare cases, acute renal failure. There is a transient increase in serum creatinine within 10 days of dosing in 1.8% of zoledronic-acid treated patients versus 0.8% of placebo-treated patients. Renal function is being monitored closely in both DATA-2 and DATA-2-EX and patients will be required to have an estimated GFR >50 (mL/min) to receive zoledronic acid 5mg. Subjects with GFR 35-50 would receive zoledronic acid 2 mg. As per the approved product labeling, the infusion time for zoledronic acid will be at least 15 minutes and will be followed by a 10 mL normal saline flush of the intravenous line.

Hypocalcemia: In clinical trials of zoledronic acid without Vitamin D pre-treatment, approximately 0.2% of patients had notable declines of serum calcium levels to values less than 7.5 mg/dL after each zoledronic acid administration. No symptomatic cases of hypocalcemia were observed in clinical trials

if they had been pretreated with Vitamin D. All patients in DATA-2-EX are being treated with Vitamin D and Vitamin D levels are being monitored in both DATA-2 and DATA-2-EX. Patients are required to have a pre-treatment 25-(OH) Vitamin-D level ≥20 (ng/mL). Patients who are administered the renal dose of zoledronic acid (2mg) will be asked to return for bloodwork 10 days (+/- 3 days) post-infusion to assess calcium and creatinine levels.

Osteonecrosis of the Jaw: Osteonecrosis of the jaw is an extremely rare side effect of zoledronic acid when given at the doses recommended for osteoporosis treatment. Subjects will not be enrolled in DATA-2-EX if they have any major dental work planned during the projected course of the study (extractions or implants). An oral examination will be performed by a study doctor prior to administration of zoledronic acid.

Atypical Femur Fractures: Atypical, low-energy, or low trauma fractures of the femoral shaft have been reported in bisphosphonate-treated patients. Atypical femur fractures may be unilateral or bilateral and some patients report prodromal dull or aching pain in the thigh in the weeks to months before a complete fracture occurs. The incidence of atypical femur fractures is not well-defined but appears to be extremely rare and at least somewhat dose-dependent. If a study subject presents with thigh or groin pain, she will be immediately evaluated to rule out an incomplete femur fracture.

#### Imaging studies

Over the 15-month study period, subjects will receive the following imaging studies:

| Study Type | DATA-2 | DATA-2-EX | Radiation |
|-------------------------------|--------------|-----------|--------------|
| | | | exposure per |
| | | | <u>scan</u> |
| DXA of the lumbar spine, hip, | 5 (including | 2 | 1 mrem |
| and radius. | screen) | | |
| HR-pQCT of the distal tibia | 4 | 2 | <0.5 mrem |
| and radius | | | |
| QCT of the hip and spine | 2 | 1 | 510 mrem |

The total dose for the DATA-2 15-month study is therefore ~1000 mrem. The total dose for DATA-2-EX (months 15-42) is ~500 mrem. This amount of radiation is equal to the background radiation one is exposed from the earth and sky over 3.25 years (for DATA-2) and 1.5 years (for DATA-2-EX).

The total dose for the observational visit alone is 0.05 mSv, equal to background radiation one is exposed from the earth and sky over 3 days.

## **VIII. Potential Benefits**

The medications given in this study have been shown to reduce fracture risk as well or better than all other approved osteoporosis therapies and subjects can expect to derive the benefit from these medications. It is hoped that the knowledge gained from this study will improve osteoporosis care.

#### IX. Monitoring and Quality Assurance

A study physician will review all laboratory test results. Subjects will be discontinued from the study if they have any finding that in the opinion of the study physician requires withdrawal from the study. Disqualifying findings will be communicated to both the subject and her primary care physician. If the subject does not have a primary care physician, the principal investigator will coordinate appropriate follow-up with a physician of the subject's choosing. Hypercalcemia is a well-described complication of teriparatide treatment. Elevated blood calcium levels will be handled in the manner recently

recommended by Antoniucci et al (see below) 57.



If serum calcium concentration is above 11.2 mg/dl, teriparatide will be stopped and serum calcium measured at least daily until normal. Thereafter teriparatide will be resumed every other day and the above algorithm followed, starting at "Reduce PTH to every other day".

The Data Safety Monitoring Board (DSMB) that is currently monitoring DATA 1 will monitor DATA 2. This DSMB is comprised of experienced clinical investigators: Dr. Deborah Wexler (Chair), Dr. Carl Pallais, and Douglass Hayden (biostatistician). Adverse events and serious adverse events will be reported to all appropriate regulatory bodies as required by current regulations.

A NIAMS-appointed DSMB will provide safety oversight for DATA-2-EX. This DSMB will meet as per NIAMS/KAI guidelines. As per NIAMS reporting requirements, all adverse events will be reported in the routine safety reports and all serious adverse events regardless of relatedness will be reported to the DSMB Safety Officer and the NIAMS, through KAI (NIAMS Executive Secretary), within 48 hours of the PI receiving notification of the events.

Adverse events or other unanticipated problems will be reported to the Partners Human Research Committee (PHRC) within 7 calendar days/5 working days of the date the investigator first becomes aware of the problem as described in the PHRC policy on Adverse Event Reporting and Unanticipated Problems Involving Risks to Subjects or Others.

#### REFERENCES

- 1. Bone health and osteoporosis: A report of the Surgeon General. In: United States Department of Health and Human Services PHS, ed.: Office of the Surgeon General; 2004.
- 2. Cummings SR, Melton LJ. Epidemiology and outcomes of osteoporotic fractures. Lancet 2002;359:1761-7.
- 3. Bliuc D, Nguyen ND, Milch VE, Nguyen TV, Eisman JA, Center JR. Mortality risk associated with low-trauma osteoporotic fracture and subsequent fracture in men and women. Jama 2009;301:513-21.
- 4. Papapoulos SE. Use of bisphosphonates in the management of postmenopausal osteoporosis. Annals of the New York Academy of Sciences 2011;1218:15-32.
- 5. Cosman F. Parathyroid hormone treatment for osteoporosis. Current opinion in endocrinology, diabetes, and obesity 2008;15:495-501.
- 6. MacLean C, Newberry S, Maglione M, et al. Systematic review: comparative effectiveness of treatments to prevent fractures in men and women with low bone density or osteoporosis. Annals of internal medicine 2008;148:197-213.
- 7. Dempster DW, Zhou H, Recker RR, et al. Skeletal histomorphometry in subjects on teriparatide or zoledronic acid therapy (SHOTZ) study: a randomized controlled trial. The Journal of clinical endocrinology and metabolism 2012;97:2799-808.
- 8. Ma YL, Marin F, Stepan J, et al. Comparative effects of teriparatide and strontium ranelate in the periosteum of iliac crest biopsies in postmenopausal women with osteoporosis. Bone 2011;48:972-8.
- 9. Stepan JJ, Burr DB, Li J, et al. Histomorphometric changes by teriparatide in alendronate-pretreated women with osteoporosis. Osteoporosis international: a journal established as result of cooperation between the European Foundation for Osteoporosis and the National Osteoporosis Foundation of the USA 2010;21:2027-36.
- 10. Dobnig H, Stepan JJ, Burr DB, et al. Teriparatide reduces bone microdamage accumulation in postmenopausal women previously treated with alendronate. J Bone Miner Res 2009;24:1998-2006.
- 11. Recker RR, Marin F, Ish-Shalom S, et al. Comparative effects of teriparatide and strontium ranelate on bone biopsies and biochemical markers of bone turnover in postmenopausal women with osteoporosis. J Bone Miner Res 2009;24:1358-68.
- 12. Jobke B, Pfeifer M, Minne HW. Teriparatide following bisphosphonates: initial and long-term effects on microarchitecture and bone remodeling at the human iliac crest. Connect Tissue Res 2009;50:46-54.
- 13. Neer RM, Arnaud CD, Zanchetta JR, et al. Effect of parathyroid hormone (1-34) on fractures and bone mineral density in postmenopausal women with osteoporosis. The New England journal of medicine 2001;344:1434-41.
- 14. Chen P, Satterwhite JH, Licata AA, et al. Early changes in biochemical markers of bone formation predict BMD response to teriparatide in postmenopausal women with osteoporosis. J Bone Miner Res 2005;20:962-70.
- 15. Ste-Marie LG, Schwartz SL, Hossain A, Desaiah D, Gaich GA. Effect of teriparatide [rhPTH(1-34)] on BMD when given to postmenopausal women receiving hormone replacement therapy. J Bone Miner Res 2006;21:283-91.
- 16. Orwoll ES, Scheele WH, Paul S, et al. The effect of teriparatide [human parathyroid hormone (1-34)] therapy on bone density in men with osteoporosis. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2003;18:9-17.

- 17. Ma YL, Zeng Q, Donley DW, et al. Teriparatide increases bone formation in modeling and remodeling osteons and enhances IGF-II immunoreactivity in postmenopausal women with osteoporosis. J Bone Miner Res 2006;21:855-64.
- 18. Keaveny TM, McClung MR, Wan X, Kopperdahl DL, Mitlak BH, Krohn K. Femoral strength in osteoporotic women treated with teriparatide or alendronate. Bone 2012;50:165-70.
- 19. Fox J, Miller MA, Newman MK, Recker RR, Turner CH, Smith SY. Effects of daily treatment with parathyroid hormone 1-84 for 16 months on density, architecture and biomechanical properties of cortical bone in adult ovariectomized rhesus monkeys. Bone 2007;41:321-30.
- 20. Compston J. The use of combination therapy in the treatment of postmenopausal osteoporosis. Endocrine 2012;41:11-8.
- 21. Pinkerton JV, Dalkin AC. Combination therapy for treatment of osteoporosis: A review. Am J Obstet Gynecol 2007;197:559-65.
- 22. Black DM, Greenspan SL, Ensrud KE, et al. The effects of parathyroid hormone and alendronate alone or in combination in postmenopausal osteoporosis. The New England journal of medicine 2003;349:1207-15.
- 23. Finkelstein JS, Wyland JJ, Lee H, Neer RM. Effects of teriparatide, alendronate, or both in women with postmenopausal osteoporosis. J Clin Endocrinol Metab 2010;95:1838-45.
- 24. Finkelstein JS, Hayes A, Hunzelman JL, Wyland JJ, Lee H, Neer RM. The effects of parathyroid hormone, alendronate, or both in men with osteoporosis. N Engl J Med 2003;349:1216-26.
- 25. Finkelstein JS, Leder BZ, Burnett SM, et al. Effects of teriparatide, alendronate, or both on bone turnover in osteoporotic men. The Journal of clinical endocrinology and metabolism 2006;91:2882-7.
- 26. Cosman F, Eriksen EF, Recknor C, et al. Effects of intravenous zoledronic acid plus subcutaneous teriparatide [rhPTH(1-34)] in postmenopausal osteoporosis. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2011;26:503-11.
- 27. Cusano NE, Bilezikian JP. Combination antiresorptive and osteoanabolic therapy for osteoporosis: we are not there yet. Curr Med Res Opin 2011;27:1705-7.
- 28. Bilezikian JP. Combination anabolic and antiresorptive therapy for osteoporosis: opening the anabolic window. Curr Osteoporos Rep 2008;6:24-30.
- 29. Valenta A, Roschger P, Fratzl-Zelman N, et al. Combined treatment with PTH (1-34) and OPG increases bone volume and uniformity of mineralization in aged ovariectomized rats. Bone 2005;37:87-95.
- 30. Kostenuik PJ, Capparelli C, Morony S, et al. OPG and PTH-(1-34) have additive effects on bone density and mechanical strength in osteopenic ovariectomized rats. Endocrinology 2001;142:4295-304.
- 31. Dempster DW, Lambing CL, Kostenuik PJ, Grauer A. Role of RANK ligand and denosumab, a targeted RANK ligand inhibitor, in bone health and osteoporosis: a review of preclinical and clinical data. Clin Ther 2012;34:521-36.
- 32. Lacey DL, Timms E, Tan HL, et al. Osteoprotegerin ligand is a cytokine that regulates osteoclast differentiation and activation. Cell 1998;93:165-76.
- 33. Yasuda H, Shima N, Nakagawa N, et al. Osteoclast differentiation factor is a ligand for osteoprotegerin/osteoclastogenesis-inhibitory factor and is identical to TRANCE/RANKL. Proc Natl Acad Sci U S A 1998;95:3597-602.
- 34. Brown JP, Prince RL, Deal C, et al. Comparison of the Effect of Denosumab and Alendronate on Bone Mineral Density and Biochemical Markers of Bone Turnover in Postmenopausal Women With Low Bone Mass: A Randomized, Blinded, Phase 3 Trial. J Bone Miner Res 2009:1-34.
- 35. Brown JP, Prince RL, Deal C, et al. Comparison of the effect of denosumab and alendronate on BMD and biochemical markers of bone turnover in postmenopausal women with low bone mass: a

- randomized, blinded, phase 3 trial. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2009;24:153-61.
- 36. Reid IR, Miller PD, Brown JP, et al. Effects of denosumab on bone histomorphometry: the FREEDOM and STAND studies. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2010;25:2256-65.
- 37. Simon JA, Recknor C, Moffett AH, Jr., et al. Impact of denosumab on the peripheral skeleton of postmenopausal women with osteoporosis: bone density, mass, and strength of the radius, and wrist fracture. Menopause 2012.
- 38. McClung MR, Lewiecki EM, Geller ML, et al. Effect of denosumab on bone mineral density and biochemical markers of bone turnover: 8-year results of a phase 2 clinical trial. Osteoporos Int 2012.
- 39. McClung MR, Zanchetta JR, Hoiseth A, et al. Denosumab Densitometric Changes Assessed by Quantitative Computed Tomography at the Spine and Hip in Postmenopausal Women With Osteoporosis. J Clin Densitom 2012.
- 40. Bolognese MA, Teglbjaerg CS, Zanchetta JR, et al. Denosumab Significantly Increases DXA BMD at Both Trabecular and Cortical Sites: Results From the FREEDOM Study. J Clin Densitom 2012.
- 41. Miller PD, Wagman RB, Peacock M, et al. Effect of denosumab on bone mineral density and biochemical markers of bone turnover: six-year results of a phase 2 clinical trial. The Journal of clinical endocrinology and metabolism 2011;96:394-402.
- 42. Bone HG, Bolognese MA, Yuen CK, et al. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women. The Journal of clinical endocrinology and metabolism 2008;93:2149-57.
- 43. Seeman E, Delmas PD, Hanley DA, et al. Microarchitectural deterioration of cortical and trabecular bone: differing effects of denosumab and alendronate. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2010;25:1886-94.
- 44. Cummings SR, San Martin J, McClung MR, et al. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med 2009;361:756-65.
- 45. Leder BZ, Tsai JN, Uihlein AV, et al. Two Years of Denosumab and Teriparatide Administration in Postmenopausal Women with Osteoporosis (The DATA Extension Study): a Randomized Controlled Trial. J Clin Endocrinol Metab 2014;jc20134440.
- 46. Tsai JN, Uihlein AV, Lee H, et al. Teriparatide and denosumab, alone or combined, in women with postmenopausal osteoporosis: the DATA study randomised trial. Lancet 2013.
- 47. Muschitz C, Kocijan R, Fahrleitner-Pammer A, et al. Overlapping and Continued Alendronate or Raloxifene Administration in Patients on Teriparatide: Effects on Areal and Volumetric Bone Mineral Density The CONFORS Study. J Bone Miner Res 2014.
- 48. Muschitz C, Kocijan R, Fahrleitner-Pammer A, Lung S, Resch H. Antiresorptives overlapping ongoing teriparatide treatment result in additional increases in bone mineral density. J Bone Miner Res 2013;28:196-205.
- 49. Leder BZ, Neer RM, Wyland JJ, Lee HW, Burnett-Bowie SM, Finkelstein JS. Effects of teriparatide treatment and discontinuation in postmenopausal women and eugonadal men with osteoporosis. The Journal of clinical endocrinology and metabolism 2009;94:2915-21.
- 50. Miller PD, Bolognese MA, Lewiecki EM, et al. Effect of denosumab on bone density and turnover in postmenopausal women with low bone mass after long-term continued, discontinued, and restarting of therapy: a randomized blinded phase 2 clinical trial. Bone 2008;43:222-9.
- 51. Black DM, Delmas PD, Eastell R, et al. Once-yearly zoledronic acid for treatment of postmenopausal osteoporosis. The New England journal of medicine 2007;356:1809-22.

15

- 52. Bolland MJ, Grey AB, Horne AM, et al. Effects of intravenous zoledronate on bone turnover and BMD persist for at least 24 months. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2008;23:1304-8.
- 53. Grey A, Bolland M, Wattie D, Horne A, Gamble G, Reid IR. Prolonged antiresorptive activity of zoledronate: a randomized, controlled trial. Journal of bone and mineral research: the official journal of the American Society for Bone and Mineral Research 2010;25:2251-5.
- 54. Grey A, Bolland MJ, Horne A, et al. Five years of anti-resorptive activity after a single dose of zoledronate--results from a randomized double-blind placebo-controlled trial. Bone 2012;50:1389-93.
- 55. Grey A, Bolland MJ, Wattie D, Horne A, Gamble G, Reid IR. The antiresorptive effects of a single dose of zoledronate persist for two years: a randomized, placebo-controlled trial in osteopenic postmenopausal women. The Journal of clinical endocrinology and metabolism 2009;94:538-44.
- 56. Reid IR, Black DM, Eastell R, et al. Reduction in the risk of clinical fractures after a single dose of zoledronic Acid 5 milligrams. The Journal of clinical endocrinology and metabolism 2013;98:557-63.
- 57. Antoniucci DM, Sellmeyer DE, Bilezikian JP, et al. Elevations in serum and urinary calcium with parathyroid hormone (1-84) with and without alendronate for osteoporosis. J Clin Endocrinol Metab 2007;92:942-7.